CLINICAL TRIAL: NCT06369519
Title: Optimization of Management for Sporadic Bilateral Renal Cell Carcinoma: a Population-based Cohort Study
Brief Title: Optimization of Management for Sporadic Bilateral Renal Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, GONG Kan, Chief physician, Peking University First Hospital
Other Study IDs: 2023#17-23
Record Dates: First submitted 2024-04-10; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Kidney Cancer
Keywords: Bilateral renal cell carcinoma; Surgery; Partial nephrectomy; Local tumor destruction; Nomogram
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Synchronous BRCC patients: Synchronous BRCC is defined as the second primary RCC emerges within 6 months from the diagnosis of the first primary RCC.
  Interventions: Procedure: Surgery treatment or local tumor destruction.
- Metachronous BRCC patients: Metachronous BRCC develops beyond 6 months from the diagnosis of the first primary RCC.
  Interventions: Procedure: Surgery treatment or local tumor destruction.

INTERVENTIONS:
Procedure: Surgery treatment or local tumor destruction. — Surgery treatments mainly include partial nephrectomy and radical nephrectomy. Local tumor destruction mainly includes renal mass ablation.

SUMMARY:
Sporadic bilateral renal cell carcinoma (BRCC) is a rare situation of RCC. The treatment for BRCC is controversial and there is a lack of authoritative guidelines about the management of BRCC. The goal of this cohort study is to identify prognostic factors, construct predictive nomograms, and optimize management for sporadic BRCC patients. The main questions it aims to answer are:

What are the factors influencing the prognosis of BRCC patients? What's the appropriate treatment for BRCC patients?

Researchers will analysis the prognostic factors and compare the prognosis of BRCC patients receiving different treatments.

DETAILED DESCRIPTION:
Sporadic bilateral renal cell carcinoma (BRCC) is a rare situation of RCC. The treatment for BRCC is controversial and there is a lack of authoritative guidelines about the management of BRCC. This cohort study aims to identify prognostic factors, construct predictive nomograms, and optimize surgical treatment for sporadic BRCC patients. The main questions it aims to answer are:

What are the factors influencing the prognosis of BRCC patients? What's the appropriate treatment for BRCC patients? In this retrospective population-based cohort study, patients diagnosed with sporadic BRCC between 2000 and 2020 were identified from the Surveillance, Epidemiology, and End Results (SEER) database. Researchers will analysis the prognostic factors and compare the prognosis of BRCC patients receiving different treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Clinical diagnosis of localized BRCC (M0) from 2000 to 2020.
* Active follow-up.
* Complete clinicopathological information.

Exclusion Criteria:

* Diagnosed by autopsy or death certificate only.
* Tending to suffer from hereditary RCC, including those complicating with pancreatic neuroendocrine tumor (pNET) or hemangioblastoma.
* Unavailable key information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was based on the Surveillance, Epidemiology, and End Results (SEER) database, which contains the population-based data from 17 Registries covering approximately 26.5% of the U.S. population. The eligible sporadic localized BRCC patients were identified from the SEER database.
Sampling Method: Non-Probability Sample
Enrollment: 3677 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | From date of diagnosis of the second primary RCC until the date of death from any cause or the date of last follow-up, whichever came first, assessed up to 20 years.
  OS was calculated as the time interval from the diagnosis of the second primary RCC to death or the time to the last follow-up.

SECONDARY OUTCOMES:
Cancer-specific survival (CSS) | From date of diagnosis of the second primary RCC until the date of death from the same disease or the date of last follow-up, whichever came first, assessed up to 20 years.
  CSS was calculated as the time interval from the diagnosis of the second primary RCC to death from the same disease or the last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Kan Gong, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Deng R, Qiu J, Shang J, Yu C, Tian P, Zhao Z, Cai L, Zhou J, Gong K. The long-term survival outcome of sporadic bilateral renal cell carcinoma and optimization of surgical treatment: a large-scale population-based cohort study. Clin Exp Med. 2024 Dec 21;25(1):20. doi: 10.1007/s10238-024-01535-5. PMID 39708253